CLINICAL TRIAL: NCT04967963
Title: Surgical Management of Stage-2 Medication-Related Osteonecrosis of the Jaw With Transplantation of Human Amniotic Membrane
Brief Title: Surgical Management of Stage-2 MRONJ With Transplantation of HAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Fatma Gülfeşan Çanakçi, Assistant Professor, Trakya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TrakyaU 2016/103
Record Dates: First submitted 2021-06-18; First posted 2021-07-20 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Medication Related Osteonecrosis of the Jaw; Oral Surgery
Keywords: Medication related osteonecrosis of the jaw; MRONJ; Amniotic membrane; Mucosal coverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transplantation of HAM (Experimental): HAM was used after sequestrectomy in patients with stage-2 MRONJ
  Interventions: Procedure: HAM

INTERVENTIONS:
Procedure: HAM — Transplantation of HAM

SUMMARY:
Medication-related osteonecrosis of the jaw (MRONJ) is a drug adverse reaction and there is no consensus for the treatment of MRONJ. The aim of this study is to evaluate the mucosal coverage using HAM after sequestrectomy in patients with stage-2 MRONJ.

DETAILED DESCRIPTION:
Medication-related osteonecrosis of the jaw (MRONJ) is a drug adverse reaction and a potentially serious complication. MRONJ is defined as the presence of exposed bone with intraoral or extraoral fistula in the maxillofacial region that does not heal for at least 8 weeks, seen in patients receiving antiresorptive or antiangiogenic agents but without a history of head and neck radiotherapy. Several treatment strategies have been recommended according to the stage of MRONJ, ranging from pharmacological conservative management to aggressive surgical approaches. According to the American Association of Oral and Maxillofacial Surgeons (AAOMS) position paper updated in 2014, conservative treatment for stage 0 and 1, minimally invasive surgical treatment for stage-2, and radical surgical treatment for stage-3 have been recommended. Furthermore, there is no consensus for the treatment of MRONJ.

The innermost membrane of the placenta; the human amniotic membrane (HAM), is an avascular membrane consisting of 5 layers: epithelium, basement membrane, compact layer, fibroblast layer, and spongy layer. HAM was used in many animal and human studies in the field of oral and maxillofacial surgery; for guided tissue regeneration, vestibuloplasty, temporomandibular joint surgery, closure of oroantral communication/fistula, periodontal surgery, oral mucosal defects, periapical endodontic surgery, cleft palate, and MRONJ.

The aim of this study is to provide mucosal coverage using HAM after sequestrectomy in patients with stage-2 MRONJ. In this case series, results of surgical treatment with HAM transplantation in 5 MRONJ cases were reported.

All donors were selected from volunteers undergoing elective cesarean section at Trakya University, Faculty of Medicine, Department of Obstetrics and Gynecology. Cryopreserved HAM was prepared as described previously by Kar et al. After preoperative clinical and radiographic evaluations, 14 MRONJ cases with stage-2 diagnosis were treated with HAM transplantation. Preoperative pain was evaluated by Visual Analogue Scale (VAS) from "0" (as no pain) to "10" (as the most severe pain experienced).

Before surgery, patients were treated with combined oral antibiotics (amoxicillin/clavulanic acid 1,000 mg + metronidazole 500 mg), oral analgesics (dexketoprofen 25 mg) and, antimicrobial mouth rinse (0.2% chlorhexidine digluconate) for 3 weeks. Surgical treatment was performed in patients who still had an infection (pain, erythema, or purulent discharge) and pain despite the medical treatment.

Surgical Method HAM was removed from the -80 °C freezer half an hour before the operation. 4% articaine hydrochloride with 1:100 000 adrenalin was used for anesthesia. Sequestrectomy was performed until fresh bleeding from bone was confirmed, with a flapless approach or a minimal flap elevation. After the sequestrectomy was completed, the amniotic membrane was placed in two layers. The deep layer HAM was placed to cover the bone surface. The superficial layer HAM was sutured with a resorbable suture (4.0 polyglactin) to the edges of the mucosa to cover the underlying bone completely. All bone specimens were histopathologically evaluated to exclude a metastatic bone malignancy or a primary malignancy of jaws. The medications described before were prescribed for 1 week.

In the first postoperative follow-up period, patients were evaluated in terms of infection (pain, erythema, and purulent drainage), mucosal coverage, and post-operative pain at 1, 2, 4, 8, and 12 weeks. Patients who showed improvement (total mucosal coverage, no sign of infection and pain) at the end of 12 weeks were followed up every 8 weeks. Also, radiographic examinations (panoramic radiography at every 8 weeks and cone-beam computed tomography at every 6 months) were performed to evaluate the progression of bone destruction postoperatively.

ELIGIBILITY:
Inclusion Criteria:

For Donors:

* Free of infections such as HIV, hepatitis B and C, and syphilis before and 6 months after the cesarean section
* Volunteers over the age of 18

For Recipients:

• Medication-related osteonecrosis of the jaw cases with stage-2 diagnosis

Exclusion Criteria:

For Donors:

* Any infection described above.
* Mentally retarded individuals

For Recipients:

* MRONJ cases with stage-1, and stage-3 diagnosis
* Mentally retarded individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in mucosal coverage | 12 weeks
  Mucosal coverage will be evaluated as "+++" for complete mucosal coverage, "++" for >50% of mucosal coverage, "+" for <50% of mucosal coverage, "-" for no improvement.

SECONDARY OUTCOMES:
Change in Pain | 12 weeks
  Pain will be evaluated by Visual Analogue Scale (VAS) from "0" (as no pain) to "10" (as the most severe pain experienced).The patient will be asked to indicate their level of on the VAS.
Change in suppuration and erythema as signs of infection | 12 weeks
  Suppuration will be evaluated as "-" is absent and "+" is present.

CONTACTS AND LOCATIONS:
Overall Officials: F. Gülfeşan Çanakçi, Study Director — Trakya University, Faculty of Dentistry
Locations (1):
- Trakya University, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Canakci FG, Er N, Duygu G, Varol GF. Surgical management of stage-2 medication-related osteonecrosis of the jaw with transplantation of human amniotic membrane: Preliminary results. J Stomatol Oral Maxillofac Surg. 2022 Jun;123(3):e28-e31. doi: 10.1016/j.jormas.2021.09.011. Epub 2021 Sep 23. PMID 34563730